CLINICAL TRIAL: NCT01110148
Title: Use of MP3 Portable Technology in Patient Education and Informed Consent of Shave and Punch Biopsies
Brief Title: Use of Portable Technology in Patient Education of Shave/Punch Biopsies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: April Armstrong, M.D., University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 200917169-1
Record Dates: First submitted 2010-04-13; First posted 2010-04-26 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Biopsy
Keywords: skin biopsy; informed consent; patient education; video education; patients requiring skin biopsies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video-based informed consent (Experimental): patients receiving informed consent through video format
  Interventions: Other: video-based informed consent for skin biopsies
- traditional informed consent (Active Comparator): patients receiving traditional informed consent from the physicians.
  Interventions: Other: traditional informed consent

INTERVENTIONS:
Other: video-based informed consent for skin biopsies — video-based informed consent for punch and shave biopsies
  Arms: Video-based informed consent
Other: traditional informed consent — traditional informed consent (standard of care) from physicians for shave and punch biopsies
  Arms: traditional informed consent

SUMMARY:
The investigators investigated the use of portable MP3 technology in patient education and informed consent of shave and punch biopsies. Eighty patients were divided randomly into a control and experimental group. Control patients received the standard of care in patient education and informed consent. Experimental patients watched a short 80-second video on shave or punch biopsies. All patients were given pre- and post-education questionnaires to assess the efficacy of each method.

ELIGIBILITY:
Inclusion Criteria:

* English speaker
* Receiving shave or punch biopsy

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Measure the post-education knowledge of each intervention arm | at the end of the study visit
  Compare the post-education knowledge between the two intervention arms: one conventional informed consent process, the other video-based informed consent process. Knowledge will be measured through a questionnaire administered before and after patient education is given.

CONTACTS AND LOCATIONS:
Overall Officials: April W Armstrong, M.D., Principal Investigator — UC Davis Health System
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States